CLINICAL TRIAL: NCT06009068
Title: Reliability and Validity of the Surgimap Software for Measuring Quadriceps Angle in Healthy Subjects
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aida Amir Nassif Naguib, Lecturer, Cairo University
Other Study IDs: P.T.REC/012/004538
Record Dates: First submitted 2023-08-19; First posted 2023-08-24 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Reliability and Validity
Keywords: Surgimap; Q-angle

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Surgimap soft ware — 20 healthy subjects will be recruited in the study, the q angle will be measured using goniometer and surgimap soft ware, 3 examiners will measure the q angles for the same individuals to check the inter rater reliability, and the test will be repeated after 2 days by the same examiners to check the intra rater reliability

SUMMARY:
The purpose of this study is to investigate the intra- and inter-rater reliability and concurrent validity of surgimap software for measuring the Q angle Surgimap (Nemaris Inc, New York, NY, USA) is a dedicated spine measurement and surgical planning software which is used in both the research works and the clinical rehabilitation. Q angle is considered to be an index of the vector for action of the patellar tendon and extensors mechanism which is highly affects the patellofemoral joint dysfunction and foot mechanics.

DETAILED DESCRIPTION:
specialised software for assessing the sagittal plane has arisen. Digital measuring software of many types has been proved to be faster, more accurate, more precise, and less variable than manual procedures. Angle measurement software is available in different formats and applications. Surgimap is another programme used for measuring angles. The current software has proven to be a godsend and is currently being used in the medical industry to measure joint angles especially the spine alignment. The programme is also used for scientific reasons, such as digital photo analysis. A recent study discovered that Surgimap software is a viable approach for evaluating spinal postural angles in teenagers from varied standing position perspectives using digital pictures.

As there a lack of knowledge about the reliability and validity of the surgimap software to measure the Q- angle. Therefore, The study will investigate the inter-rater, intra-rater reliability and concurrent validity of the surgimap software for measuring the Q-angle.

ELIGIBILITY:
Inclusion Criteria:

* Both male & female
* Aged 18:25
* BMI 18.5: 25
* Normal foot posture as assessed by foot posture index.

Exclusion Criteria:

* Subjects who have operations in the knee joint
* Subjects who have traumatic knee injury
* High arched or low arched foot.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: This study will be conducted in the out-patient clinic Faculty of physical therapy, Cairo University. The expected duration to recruit patients and collect data is 3 months .
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-08-30 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
The inter-rater, intra-rater reliability and concurrent validity of the surgimap software for measuring the Q-angle. | 3 months
  the accuracy and consistency of surgimap software for measuring the q angle

CONTACTS AND LOCATIONS:
Overall Officials: Aida Nassif, PHD, Principal Investigator — lecturer of physical therapy, Cairo University
Locations (1):
- Faculty of physical therapy, Cairo University, Giza, Egypt